CLINICAL TRIAL: NCT00139516
Title: Chinese Community Smoking Cessation Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 247; R01HL069363 (NIH)
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Lung Diseases; Diabetes Mellitus; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Lung Diseases; Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive | interventions — Nicotine Replacement Therapy

INTERVENTIONS:
Behavioral: self-help
Drug: nicotine replacement therapy
Behavioral: smoking cessation

SUMMARY:
The study has two objectives/aims:

Aim 1: To test the efficacy of the intervention among adult smokers with cardiovascular disease, pulmonary disease and diabetes mellitus related illnesses (later modified to Chinese adults with and without diseases); and

Aim 2: To examine a set of measures (background, general health, psychosocial, and smoking process) that are associated with smoking cessation at 6 and 12 months

DETAILED DESCRIPTION:
BACKGROUND:

Studies of smoking cessation intervention among hospitalized patients with CVD and pulmonary disease produced varying cessation rates, ranging from 20 to 51% among patients with pulmonary disease, from 22 to 71% among survivors of coronary disease and as much as 80% among lung cancer patients (3-8). Recently published Treating Tobacco Use and Dependence Clinical Practice Guideline (1) provides detailed evaluation and synthesis of evidence-based components of effective smoking cessation interventions and summary results for selected treatment modalities are presented in Table 1. Face-to-face counsel, strong advice from physician or nurse, the number of reinforcing sessions and duration of these sessions were related to success (9). Compared to no treatment, estimated abstinence rates for treatment modalities ranged from 10.2% to 26.5%. Thus, use of combination treatment modalities in smoking cessation intervention is expected to result in higher abstinence rate.

The proposed four-year prospective, randomized clinical trial with 12 months follow-up, will test the efficacy of a culturally and linguistically tailored physician directed, nurse managed, smoking cessation and relapse prevention intervention among Chinese smokers. The study has two aims: 1) To test the efficacy of the intervention among smokers; and 2) To examine a set of measures (background, general health, psychosocial, and smoking process) that are associated with smoking cessation at 6 and 12 months. Subjects who smoked in the 3 months prior to admission at 6 San Francisco Bay Area hospitals (1 university, 4 private and 1 county) will be screened, recruited and randomized to one of two interventions: a) Intensive [n=190] (physician advice, bedside counseling with a family member, 5 telephone contacts within 90 days, with nicotine replacement therapy and one repeat relapse counseling with 1 more telephone contact for relapsers). b) Minimal [n=190] (physician advice and a self-help manual). Random assignment will be stratified by recruitment site, gender and disease category. Primary outcomes include biochemically confirmed abstinence and quit attempts at 6 and 12 months. Power calculation is based on 15% difference in abstinence rates between the two intervention groups. The findings from this propose study will yield significant knowledge for effectively treating Chinese smokers and will provide insight into treatment for smokers of other racial and ethnic minorities that is likely to have significant public health impact by reducing health disparities among US sub-populations.

DESIGN NARRATIVE:

A prospective, randomized clinical trial with 12-month follow-up linguistically tailored, nurse-managed smoking cessation and relapse prevention trial. It involves several stages in the study:

Stage 1: Recruitment - verify eligibility criteria and making phone appointment for face-to-face baseline interview and individualized counseling session.

Stage 2: Baseline face-to-face interview either in a hospital setting for inpatients, or in an office setting for those who were not inpatients - explain study, obtained informed consent, conducting baseline survey and randomized patients into one of two research arms: Intensive or minimal. Intensive patients will receive a specific set of interventions and asked to contract a quit date, whereas minimal subjects will receive the usual care and advice to quit from the research staff and their physicians.

Stage 3: For subjects randomized to the intensive group, they will receive a set of intervention support phone calls for their quit-smoking efforts.

Stage 4: Outcome Measurement - All subjects will receive 6- and 12-month phone calls and saliva samples will be collected to verify non-smoking status. At six months - interim outcome, at 12 months - final outcome measurement.

Procedures

Cognitive Pretest:

We conducted pretest of the translated materials using individual interviews to ascertain their face validity. Participants for the cognitive pretest were either bilingual or fluent in either English or Chinese. These participants will include both current and recent ex-smokers from the community who speak either Mandarin or Cantonese (the two most commonly spoken Chinese dialects).

Intervention:

Participants assigned to the minimal intervention group will receive physician advice and a standard self-help manual, either an English version of "Freedom From Smoking" from the American Lung Association (ALA), or a Chinese version "Victory over Smoking," (see attached). The physician advice consists of a strong message urging the patient to quit smoking (see attached). Physicians will be prompted to deliver a 1- to 2-minute unequivocal scripted message about the necessity to quit smoking. For the inpatients, a 1-page prototype Physician Advice Statement will be placed in the progress notes section of the patient's medical record to serve as a physician reminder. For the outpatients, if the first counseling session is done outside of the physician's office setting, the 1-page prototype will be faxed to the physician's office to notify the physician and to remind them to counsel the study subjects. If the counseling is done in the physician's office, the 1-page prototype will be given directly to the patients physician or be placed inside the office chart in his absence.

Participants in the intensive group will receive the nurse- or health educator-managed smoking cessation and relapse prevention intervention. The intensive intervention has two periods: initial counseling session and follow-up phone support.

Initial Counseling Session - Patients in the intensive group will receive the scripted physician advice as well as an endorsement from their physicians about the nurse/health educator-managed smoking cessation intervention. A nurse/health educator-mediated behavioral counseling will be provided after obtaining the baseline smoking history and determining self-efficacy for smoking cessation. The 60- to 90-minute nurse/patient educator-managed intervention includes components of patient education, skill building and relapse prevention counseling. During this session, the patient will be given individually-tailored counseling based on his/her baseline assessment information. They will also be given a 20-minute smoking cessation video in Chinese, a Chinese workbook Victory over Smoking self-help manual, based on the Freedom From Smoking workbook from the American Lung Association, and a 15-minute relaxation audiotape in Chinese.

Although the primary focus of the intervention is a cognitive behavioral intervention, nicotine replacement therapy (NRT) will be offered to patients who do not have medical contraindications to the NRT and: a) meet the criteria for nicotine dependency; or b) are noted by the nurses to have severe withdrawal symptoms (inpatients) or self-report severe withdrawal symptoms during previous quit attempts,; c) relapse after the initial counseling; and d) smoke more than 10 cigarettes a day.

For patients in either group who have been smoking within the 7 days prior to the time of the interview, 2-3 cc of saliva will be collected from them for studying the metabolic rate of cotinine.

Patients will be offered NRT by trained nurse/health educators, in the form of gum (Nicorette 2 or 4 mg) or patch (Nicoderm 14 or 21 mg), depending on patients' preference. We will obtain the approval from each subject's physician before providing NRT. Upon physician consent, patients will be instructed in the correct use of nicotine patch or gum by nurses/health educators using an 8-week protocol for both the nicotine patch and gum) [see NRT protocol].

Post-Counseling Period (from 2 to 90 days) - During this period, the nurses/health educators will contact patients in the intensive group beginning 48 hours post discharge for the inpatients, and 48 hours post patients' quit dates for the outpatients. Additional calls are made at 7-, 21-, 45- and 90-day intervals during the period of greatest risk for relapse (9). Reinforcements for proper nutrition, physical activity and enlisting support from family members and friends will be provided during each 10-minutes telephone follow-up contact. If the subjects relapse during the first 90-day period of enrollment (identified through scheduled telephone calls by nurses/ health educators), they will be offered one additional intervention telephone call. The purpose of this call is to review the smoking cessation materials that had been originally presented to the subject, to continue problem solving with the subject regarding high-risk situations that led to relapse, and to reinforce the importance of quitting smoking permanently.

The primary focus of our intervention is in cognitive behavioral intervention. Nicotine replacement therapy is only one component of the intensive intervention. Because NRT is considered a standard of care, we are not proposing to withhold NRT but rather will not offer the medication as part of the minimal intervention. Regardless of the intervention arms, participants will be able to take NRT either on their own or as prescribed by their clinicians. The nurse/health educator will record the use of NRT among all the other participants who are treated with NRT.

Intervention Follow-up Assessments:

After the intervention, all subjects will be reassessed by scripted telephone interviews at 6 and 12 months (see attached). Each telephone call will take approximately 10 minutes. Nurses/health educators will be blinded to group assignment as they made follow-up calls. Initial questions assess smoking status and categorize each subject into one of three categories: nonsmoker (had not smoked since the initial counseling session or the last telephone call), relapser (had smoked since the initial counseling session or the last telephone call but not on a continuous basis), or continuous smoker (had smoked daily for the past 7 days). After each assessment, a saliva sample collection kit will be mailed out to the non-smoking participants with instructions and a postage-paid envelope for return. Participants who have not returned their cotinine within 15 days will be contacted by telephone.

ELIGIBILITY:
Inclusion Criteria:

* having smoked a cigarette, cigar, or tobacco pipe during the 3 months preceding the baseline interview
* reside in the San Francisco Bay Area at baseline
* must be fluent in either English or Chinese (Mandarin or Cantonese)
* be 18 and over in age and
* not currently engaging in assisted smoking cessation efforts

Exclusion criteria

* unable to speak English or Chinese
* too ill to participate, or not willing to participate in smoking cessation effort
* pregnancy
* major psychiatric illness not under control/treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candice Wong — University of California at San Francisco